CLINICAL TRIAL: NCT01644084
Title: A Comparison Between 5% Albumin and 6% Hydroxyethyl Starch 130/0.4 in Priming Solution for Cardiopulmonary Bypass and Post-bypass Maintenance Fluid in High-risk Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 4-2009-0061
Record Dates: First submitted 2012-07-16; First posted 2012-07-18 (Estimated); Last update posted 2012-07-19 (Estimated); Status verified 2012-07

CONDITIONS: Patients Undergoing Cardiac Surgery With Cardiopulmonary Bypass
Keywords: albumin; hydroxyethyl starch 130/0.4; cardiopulmonary bypass
MeSH Terms: interventions — Hydroxyethyl Starch Derivatives

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- HA (priming)-HES (up to 15 ml/kg after CPB) (Experimental)
  Interventions: Drug: Hydroxyethyl starch 130/0.4
- HES (priming)-HES (up to 15 ml/kg after CPB) (Active Comparator)
  Interventions: Drug: Hydroxyethyl starch 130/0.4
- HA (priming)-nonHES (only crystalloids after CPB) (Active Comparator)
  Interventions: Drug: Hydroxyethyl starch 130/0.4

INTERVENTIONS:
Drug: Hydroxyethyl starch 130/0.4 — Hydroxyethyl starch 130/0.4 as a priming of cardiopulmonary bypass circuit and/or as a fluid after cardiopulmonary bypass
  Arms: HA (priming)-HES (up to 15 ml/kg after CPB)
Drug: Hydroxyethyl starch 130/0.4 — Hydroxyethyl starch 130/0.4 as a priming of cardiopulmonary bypass circuit and/or as a fluid after cardiopulmonary bypass
  Arms: HES (priming)-HES (up to 15 ml/kg after CPB)
Drug: Hydroxyethyl starch 130/0.4 — Hydroxyethyl starch 130/0.4 as a priming of cardiopulmonary bypass circuit and/or as a fluid after cardiopulmonary bypass
  Arms: HA (priming)-nonHES (only crystalloids after CPB)

SUMMARY:
It is advantageous to use 5% human albumin (HA) in patients undergoing cardiopulmonary bypass (CPB), because preexposure of the synthetic surfaces of the CPB circuit to albumin decreases coagulopathy, platelet aggregation, immune responses. However the use of albumin is limited, because it is expensive and can rarely cause infection.

Hydroxyethyl starch (HES) decreases clot strength and prolong clot formation. A recently developed 6% HES 130/0.4 is known to have fewer effects on hemostasis. However Schramlo AA et al. reported that short time infusion of HES 130/0.4 after cardiac surgery produced impairment in fibrin formation and clot strength in thromboelastometry tracings.

Coagulopathy is directly related to bleeding and massive postoperative bleeding increases the risk of reoperation. Therefore it is important to avoid administration of fluids that can inhibit homeostasis after CPB.

The purpose of this study is to investigate the effect of 6% HES 130/0.4 as a component of priming solution on coagulation compared to 5% HA.

ELIGIBILITY:
Inclusion Criteria:

* patients who have uncontrolled medical problems, life-threatening cardiac disease, complex cardiac surgery, or emergency operation

Exclusion Criteria:

* patients who had received warfarin, heparin, acetylsalicylic acid, or antiplatelet drug within 5 days before surgery

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2009-06; Primary Completion 2011-01 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Effect of 6% hydroxyethyl starch 130/0.4 as a priming solution on coagulation and blood loss following complex heart valve surgery: a comparison with 5% albumin | upto 24hours after cardiopulmonary bypass
  The purspose of this study is to investigate the effect of 6% HES 130/0.4 as a component of priming solution on coagulation compared to 5% HA. Rotation thromboelastography (ROTEM) was performed before and 24 h after CPB. Hemoglobin, platelet count and transfusion requirement were assessed for 24 h postoperatively.

CONTACTS AND LOCATIONS:
Locations (1):
- Yonsei Univ. dept. of Anesthesiology and pain medicine, Seoul, Seoul, South Korea